CLINICAL TRIAL: NCT02668302
Title: The PIO II Study: A Randomized, Controlled, Blinded Trial to Evaluate the Safety and Efficacy of In-office Placement of a Steroid-eluting Sinus Implant Post-ethmoidectomy
Brief Title: The PIO II Study: In-office Post-op Placement of a Steroid-eluting Sinus Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Collin County Ear Nose & Throat (Other)
Collaborators: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P2015-09
Record Dates: First submitted 2016-01-04; First posted 2016-01-29 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Chronic Sinusitis, Ethmoidal
Keywords: Steroid-eluting sinus implant; Mometasone furoate; Endoscopic sinus surgery
MeSH Terms: interventions — Mometasone Furoate; Debridement; Therapeutic Irrigation; Steroids

STUDY DESIGN:
Intervention Model Description: Patients assigned to the treatment group underwent a bilateral in-office placement of a steroid-eluting sinus implant 7 days following ethmoidectomy in addition to post-op standard of care, including debridement, irrigation, and topical steroids. Patients randomized to the control group received same standard of care alone.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were wearing eye masked and noise-cancelling headsets during placement and follow-up endoscopies.
  The primary outcome was assessed by an independent sinus surgeon based on a centralized, blinded video-endoscopy review.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Bilateral in-office placement of a steroid-eluting sinus implant following ethmoidectomy in addition to post-op standard of care, including debridement, irrigation, and topical steroids
  Interventions: Combination Product: Steroid-eluting sinus implant; Other: Post-op standard of care
- Control (Active Comparator): Post-op standard of care, including debridement, irrigation, and topical steroids
  Interventions: Other: Post-op standard of care

INTERVENTIONS:
Combination Product: Steroid-eluting sinus implant — PROPEL (Intersect ENT, Inc., Menlo Park, CA), containing 370μg of mometasone furoate gradually released over 30 days
  Other Names: PROPEL
  Arms: Treatment
Other: Post-op standard of care — Post-op standard of care including debridement, irrigation, and/or topical steroids
  Other Names: Debridement, irrigation, topical steroids

SUMMARY:
Randomized, controlled, blinded clinical trial with 40 patients randomized in a 1:1 ratio to either treatment (bilateral in-office placement of a drug-eluting implant in the ethmoid sinuses following ethmoidectomy) or control (post-op standard of care) group and followed for 6 months.

DETAILED DESCRIPTION:
This prospective, randomized, controlled, blinded trial aimed to assess the efficacy of a drug-eluting sinus implant placed following ethmoidectomy in addition to post-op standard of care, including debridement, irrigation, and topical steroids, compared to the same standard of care alone (control). Patients returned for follow-up examination at 2 weeks and again at 1, 3 and 6 months after placement. Follow-up examination consisted of patient-reported outcomes and endoscopic grading by clinical investigators and an independent sinus surgeon based on a centralized, blinded video-endoscopy review.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic rhinosinusitis, defined by the AAO-HNS 2015 guidelines, including presence of bilateral ethmoid disease.
* ESS including bilateral ethmoidectomy with middle meatal antrostomy within 7 days prior to scheduled implant placement. Concurrent septoplasty and surgical treatment of the other paranasal sinuses also permitted.

Exclusion Criteria:

* Known history of intolerance to corticosteroids or an oral steroid-dependent condition.
* Known history of immune deficiency, insulin-dependent diabetes, cataracts, or glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith E Matheny, MD, Principal Investigator — Collin County Ear Nose & Throat
Locations (1):
- Collin County Ear Nose & Throat, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 45 patients were recruited at one clinical site between November 9, 2015 and May 24, 2016, of whom 40 met final eligibility.
Pre-assignment Details: Participants underwent endoscopic sinus surgery, including bilateral ethmoidectomy with middle meatal antrostomy. Concurrent septoplasty and surgical treatment of the other paranasal sinuses were also permitted. Participants returned at 7 days post-op and those meeting final eligibility underwent baseline assessment and group assignment.
Groups:
- Sinus Implant+Post-op Standard of Care: Bilateral in-office placement a steroid-eluting sinus implant in the ethmoid sinuses in addition to post-op standard of care, including debridement, irrigation, and topical steroids
- Post-op Standard of Care: Post-op standard of care, including debridement, irrigation, and topical steroids
Period: Overall Study
Arm/Group | Sinus Implant+Post-op Standard of Care | Post-op Standard of Care
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Treatment: Steroid-eluting sinus implant placement following ethmoidectomy in addition to post-op standard of care (i.e. debridement, irrigation, and topical steroids)
- Control: Post-op standard of care (i.e. debridement, irrigation, and topical steroids)
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (12.81) | 51.6 (10.83) | 50.1 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Number of prior ESS [Count of Participants; unit: Participants] — Prior endoscopic sinus surgery procedures
  Participants
    None | 17 | 14 | 31
    1 ESS | 1 | 4 | 5
    2 ESS | 0 | 1 | 1
    3 ESS | 1 | 0 | 1
    4 ESS | 1 | 1 | 2
History of asthma diagnosed by physician [Count of Participants; unit: Participants] | 6 | 4 | 10
History of allergic rhinitis diagnosed by physician [Count of Participants; unit: Participants] | 10 | 9 | 19
History of allergies [Count of Participants; unit: Participants]
  None | 7 | 8 | 15
  Environmental | 8 | 5 | 13
  Food | 2 | 2 | 4
  Other | 8 | 8 | 16
History of aspirin exacerbated respiratory disease (AERD) [Count of Participants; unit: Participants] | 0 | 0 | 0
History of smoking [Count of Participants; unit: Participants]
  Never smoked | 13 | 15 | 28
  Former smoker | 6 | 4 | 10
  Current smoker | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Inflammation Score
Description: Inflammation score was determined at baseline and Day 90 using a visual analogue scale (VAS), ranging from 0 (no visible inflammation) to 100 (severe inflammation, involving significant and extensive erythema and edema and/or hypertrophy and/or polypoid changes), as determined by an independent sinus surgeon based on a centralized, blinded video-endoscopy review.
Time Frame: Change from baseline to Day 90
Population: Intent-to-treat population (all randomized participants). Values adjusted for any surgical or steroid intervention by caring forward last observation before intervention. Scores for 9 participants (7 treatment, 2 control) were missing because the video-endoscopies for those participants had insufficient content to allow grading.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sinus Implant+Post-op Standard of Care | Post-op Standard of Care
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 26.7 (8.24) | 26.8 (6.27)
  Day 90: number analyzed (Participants) | 16 | 18
  Day 90 | 21.5 (20.84) | 17.6 (8.83)
  Change from baseline: number analyzed (Participants) | 13 | 18
  Change from baseline | -5.2 (24.36) | -9.7 (9.20)
Statistical Analysis 1: Comparison: Sinus Implant+Post-op Standard of Care vs Post-op Standard of Care; Test type: Superiority; p = 0.4709, t-test, 2 sided; P-values from two-sample T-test with equal variance assumption

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/20
Other Adverse Events (participants affected / at risk) | 6/20 | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=20) | Control (N=20)
Pelvic abscess (Reproductive system and breast disorders) | 1 | 0 — Patient was hospitalized for pelvic abscess following hysterectomy. The event was judged unrelated to the steroid-eluting sinus implant or placement procedure.
Myocardial Infarction (Cardiac disorders) | 1 | 0 — Participant had pre-existent cardiac disease. The event was determined to be unrelated to the steroid-eluting implant or placement procedure
Synechiae nose (Surgical and medical procedures) | 0 | 1 — Synechiae resulting from the middle turbinate lateralization requiring intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=20) | Control (N=20)
Sinusitis (Infections and infestations) | 1 | 1
Congestion chest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Participant complained of chest congestion
Congestion nasal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergy aggravated (Immune system disorders) | 0 | 1
Cellulitis nasal (Infections and infestations) | 1 | 0 — Cellulitis inside right nasal vestibule treated with antibiotics
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pain ear (Ear and labyrinth disorders) | 1 | 0 — Participant complained of ear pain. It was judged to be unrelated to the steroid-eluting sinus implant.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
* Small sample size
* Large intragroup variability
* Technical issues with video-endoscopies resulted in missing values for the primary endpoint in 7 (35%) treatment and 2 (10%) control participants, not allowing to draw any conclusions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No